CLINICAL TRIAL: NCT03026985
Title: Acute Skeletal Muscle Wasting and Relation to Physical Function in Patients Requiring Extracorporeal Membrane Oxygenation (ECMO)
Brief Title: Acute Skeletal Muscle Wasting and Relation to Physical Function in Patients Requiring ECMO
Status: Completed | Type: Observational
Sponsor: The Alfred (Other)
Responsible Party: Principal Investigator, Kate Hayes, Senior Physiotherapist, The Alfred
Other Study IDs: 516/16
Record Dates: First submitted 2017-01-15; First posted 2017-01-20 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Critical Illness; Muscle Wasting; Extracorporeal Membrane Oxygenation
Keywords: Extracorporeal Membrane Oxygenation; Ultrasonography; Intensive Care Units
MeSH Terms: conditions — Critical Illness; Muscular Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational cohort: Ultrasound measurement of quadriceps muscle size and echogenicity will be obtained at baseline (within 48 hours of ECMO commencement), 10 days and 20 days after baseline measurement.
  Measures of muscle strength and highest mobility level will be obtained at day 10 and day 20 after baseline measurement in order to determine the relationship between these volitional measures and the ultrasound parameters.
  Interventions: Other: Observational cohort

INTERVENTIONS:
Other: Observational cohort — Ultrasound assessment of quadriceps, muscle strength testing, highest mobility level

SUMMARY:
The purpose of this study is to describe the changes in quadriceps muscle size and quality over the first 10 days on extracorporeal membrane oxygenation (ECMO) using ultrasound imaging. This study will also examine the relationship between those changes and muscle strength and level of physical function at day 10 and day 20 after ECMO commencement.

DETAILED DESCRIPTION:
The use of ECMO has increased dramatically in the past decade with improvements in technology and survival. Whilst it is a potentially life-saving intervention in a group of patients at high risk of death, it is both highly invasive and expensive. ECMO poses a dramatic physiological burden on patients with major long-term consequences. Among these, severe prolonged neuromuscular weakness is perhaps the most significant complication. Described clinically as intensive care unit acquired weakness (ICUAW), it is associated with prolonged weaning from mechanical ventilation, delayed rehabilitation, increased hospital length of stay, and mortality with residual deficits in physical functional ability persisting up to 5 years following the ICU admission. The health value, to both patients and society, could be substantially improved if more patients achieved a complete recovery.

Muscle strength testing in the early stages of critical illness is limited, as it requires the patient to be awake, alert and cognitively intact, therefore delayed diagnosis of ICUAW due to inability of patients to complete muscle strength testing is common. Consequently, there is growing interest in the utility of ultrasound imaging to monitor the trajectory of muscle wasting and inform development of targeted interventions in these critically ill patients. Ultrasound imaging of skeletal muscle is a non-invasive, painless and radiation free technique that can provide objective, accurate and reliable data on skeletal muscle in these critically ill patients. This study will use ultrasound imaging to quantify the early change in skeletal muscle size and quality, and the relationship to strength and physical function in patients on ECMO. Risk stratification of patients with peripheral muscle wasting is vital for optimising clinical management, including development of improved rehabilitative strategies to improve recovery and optimise the risk/benefit profile of ECMO.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years)
* Requiring ECMO for management of severe cardiac or respiratory failure
* Likely to spend > 24 hours on ECMO

Exclusion Criteria:

* Presence of:
* Any connective tissue disorders (e.g., Marfan's syndrome)
* A proven or suspected acute primary brain process that is likely to result in global impairment of conscious level or cognition, such as traumatic brain injury, intracranial haemorrhage, stroke, or hypoxic brain injury after cardiac arrest or asphyxiation
* Any neuromuscular conditions (e.g., multiple sclerosis, muscular dystrophy, spinal cord injury, Guillain-Barre syndrome)
* Any current cancer or chemotherapy
* A cognitive impairment prior to the acute illness that is associated with admission to ICU that would impair capacity to follow verbal instructions Any current acute musculoskeletal injuries of hip, knee, and ankle
* A pre-existing mobility impairment where the patient is unable to walk without assistance prior to the acute illness that is associated with admission to ICU (use of a walking stick or frame is not an exclusion)
* A language barrier to patient comprehension, or where death is deemed imminent and inevitable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult critically ill patients admitted to the ICU requiring ECMO
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2017-09-19 (Actual); Study Completion 2017-09-19 (Actual)

PRIMARY OUTCOMES:
Change in quadriceps muscle size as determined by ultrasound in patients requiring ECMO | 10 days
  Change in quadriceps muscle size

CONTACTS AND LOCATIONS:
Overall Officials: Kate Hayes, Principal Investigator — The Alfred
Locations (1):
- Alfred Health, Melbourne, Australia

IPD SHARING:
Plan to Share IPD: No